CLINICAL TRIAL: NCT06809556
Title: Association of Processed Electroencephalography Derived Parameters with Postoperative Delirium in Patients with Parkinson's Disease Undergoing Elective Neurosurgery
Brief Title: Association of EEG Parameters with Postoperative Delirium in Patient's with Parkinson's Disease
Status: Not yet recruiting | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Sujoy Banik, Anesthesiologist, Assistant Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: POD in Parkinson's Patients
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Post Operative Delirium; Parkinson Disease
Keywords: post operative delirium; Parklinson's Disease; EEG
MeSH Terms: conditions — Emergence Delirium; Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- EEG (electroencephalogram) monitoring of Parkinson's patients undergoing deep brain stimulation: Parkinson's patients undergoing deep brain stimulation (DBS). Patients will undergo DBS according to institutional protocol and monitoring via EEG will be used to detect burst suppression signals. Patients will undergo cognitive testing via completion of the 3D CAM (3-minute diagnostic interview for confusion assessment method-defined delirium) tool within 15 minutes of arriving to the surgical recovery area after the completion of surgery, discharge from the recovery area, and 24 hours postoperatively. The patients' MoCA (Montreal Cognitive Assessment) score would also be assessed at 24 hours postoperatively.
  Interventions: Other: EEG (electroencephalogram) monitoring of Parkinson's patients undergoing deep brain stimulation

INTERVENTIONS:
Other: EEG (electroencephalogram) monitoring of Parkinson's patients undergoing deep brain stimulation — Parkinson's patients undergoing deep brain stimulation (DBS) will be monitored with EEG to detect burst suppression signals during surgery and will undergo postoperative cognitive testing for postoperative delirium.

SUMMARY:
Patients with Parkinson's disease seem prone to developing postoperative delirium after surgery, the causes of which remain understudied and multifactorial. Anesthetic management remains challenging due to the changes in neurotransmitter levels in these patients which translate to altered drug effects. Avoiding excessive anesthesia is essential. Processed electroencephalography (EEG) is used worldwide along with our centre to monitor depth of anesthesia. It is non-invasive and easy to use. Some EEG patterns like "burst suppression" are easily identifiable and indicate that the brain has fallen into an excessively low metabolic state, which could mean increased anesthetic sensitivity. Appearance of "burst suppression" can predict delirium in non-neurosurgical procedures, but this has never been studied during surgery for deep brain stimulator insertion in Parkinson's disease patients. Through this study we wish to observe the association of EEG parameters with the development of postoperative delirium in this subset of the population.This has the capacity to change anesthetic practice by being mindful of the fragile brain of such patients and individualizing drug dosing for each patient to improve outcomes and reduce hospital stay.

DETAILED DESCRIPTION:
Postoperative delirium is a multifactorial condition, with incidence ranging from 20% to 50%. Unfortunately, the implications of postoperative delirium extend beyond the immediate perioperative period. Bickel et al observed in their three-year follow-up that patients experiencing postoperative delirium (POD) exhibited cognitive decline and had an elevated risk of developing dementia compared to those without delirium after orthopedic surgeries.

Parkinson's disease is a neurodegenerative disorder that has been associated with an increased risk of developing delirium, with a prevalence rate of 34%. The incidence of postoperative delirium in this subset, reported after DBS in Parkinson's patients, ranges from approximately 22% to as high as ~43%. Patients with Parkinson's disease commonly undergo various elective surgical procedures, including deep brain stimulation (DBS) electrode insertion. The anesthetic management for DBS generally involves monitored anesthesia care with mild sedation, followed by patient awakening for microelectrode recording (MER) to ensure optimal electrode positioning. Increased propensity for postoperative delirium in these patients with Parkinson's has prompted foray into its predictive factors.

Intraoperative EEG has demonstrated significant promise as a predictor of postoperative delirium, especially in the elderly. A systematic review and meta-analysis by Likhvantsev et al found that the presence of burst suppression was associated with a 41% increase in the relative risk of POD, and the duration of burst suppression correlated with a higher occurrence of postoperative cognitive dysfunction (POCD). Presence and duration of burst suppression in the intraoperative period was found to be an independent predictor of postoperative delirium. In instances of delirium occurring in the absence of burst suppression, low absolute and relative frontal alpha power have been associated with its incidence.

Interestingly, all previous studies were conducted in patients without preexisting neurological conditions, with minimal literature focusing on intraoperative processed EEG in patients with Parkinson's. In an observational study by Astalosch et al, intraoperative burst suppression was found to be an influencer for the severity of delirium. There exists a significant gap in the evidence regarding the utility of intraoperative EEG-derived parameters in predicting the occurrence of delirium in Parkinson's disease.

Postoperative delirium, along with causing increased morbidity and longer hospital stay, could also lead to long-term effects, such as cognitive decline and increased vulnerability to dementia. And in patients with Parkinson's, due to consequence of delirium, there are reports higher mortality rate as compared to healthy individuals. Despite the recognized higher incidence of delirium and its effects in this patient population, there is a notable lack of research exploring intraoperative EEG-based predictors. This study aims to investigate the utility of presence of burst suppression, (along with various other processed EEG based parameters) as potential indicators of postoperative delirium in patients undergoing DBS. By exploring these factors, we hope to identify reliable markers of postoperative delirium that help us identify patients at risk, refine anesthetic techniques to minimize risk, ultimately enhance the quality of care provided to this particularly vulnerable set of patients.

All the patients will undergo preanesthetic evaluation as per institutional protocol and intraoperative anesthetic management will be performed as per institutional protocol. Patients' surgery and follow up care will proceed according to plan and standard of care and will not be altered due to participation in this study. Informed and written consent will be obtained.

After wheeling into the OR, monitoring will be instituted as per the Canadian Anesthesiologists' Society (CAS) standards. Processed electroencephalography will be monitored using Patient State Index (PSI, SedlineTM Masimo, USA) monitor. First stage of the procedure is performed under sedation with awake testing phase. Choice of sedative agent, its dosing and titration will be at the discretion of the treating anesthesiologist. Stage II of the procedure for implantable pulse generator (IPG) placement will be conducted under general anesthesia with endotracheal tube. Drugs used for general anesthesia, doses (boluses, infusion rates, and cumulative totals, as applicable) and duration of administration will be noted. Hemodynamic and fluid management during the intraoperative period will be as per the treating anesthesiologist.

Hemodynamic variables [heart rate (HR), systolic blood pressure (SBP), diastolic blood pressure (DBP), oxygen saturation (SpO2)] will be recorded at every 15 minutes. Number of episodes of hypertension (defined as SBP >180 mm Hg) or hypotension (defined as SBP< 90 mm Hg) will be noted. Episodes of desaturation (defined as SpO2 <92%) and treatment instituted for the same will be recorded. If any further samples are drawn (if needed by the attending anesthesiologist) for blood gas analysis in the intraoperative period, they will be noted.

Intraoperative blood loss, amount of fluid administered, and intraoperative adverse events (Hypo/hypertension/ hypoxemia/ seizure/ agitation/ delirium/ conversion to general anesthetic/ need for airway intervention/ nausea and vomiting) will be recorded. After emergence, patient will be shifted to postanesthesia care unit (PACU).

Postoperative hemodynamics and SpO2 on arrival in PACU will be recorded. Arterial sample will be collected for a repeat blood gas plus analysis in the PACU, and all parameters noted. Postoperative delirium scoring and cognitive assessment will be performed by a member of the research team. Postoperative adverse events and treatment instituted will be noted. All the interventions made by the nursing team in case of delirium will be made note of (hearing/visual aids/ analgesia/ presence of family member/ restraints use etc).

3D CAM scoring will be used to assess delirium on arrival to PACU, at discharge from PACU, and at 24 hours postoperatively. MoCA (Montreal Cognitive Assessment) score would also be assessed at 24 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Parkinson's disease
2. Elective neurosurgery for implantation of DBS electrodes and implantable pulse generator (IPG) device.
3. 18 years of age or older

Exclusion Criteria:

1. Refusal/withdrawal of consent
2. Inability to place sensor/ record EEG for the entire duration of surgery
3. Emergency surgery
4. Redo surgery
5. Preoperative delirium (defined as per 3D CAM score)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or older who have been diagnosed with Parkinson's Disease and are undergoing elective neurosurgery for implantation of DBS electrodes and implantable pulse generator (IPG) device.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Identification and quantification of the association between the presence of intraoperative burst suppression with the incidence of postoperative delirium | During surgery to 24 hours postoperative
  Identification and quantification of the association between the presence of intraoperative burst suppression with the incidence of postoperative delirium. This will be measured by evaluating the presence of burst suppression readings found during intraoperative EEG monitoring and determining whether the readings are associated with the development of postoperative delirium (measured by the administration of the 3D CAM and MoCA tools).

SECONDARY OUTCOMES:
Determining the association of postoperative delirium with other parameters on perioperative processed EEG | During surgery to 24 hours postoperative
  EEG readings will be assessed to determine if duration (minutes) of burst suppression, peak frontal alpha power, and duration (minutes) of patient state index (PSI) are associated with the development of postoperative delirium (measured by the administration of the 3D CAM and MoCA tools).

CONTACTS AND LOCATIONS:
Overall Officials: Sujoy Banik, MD, Principal Investigator — Western University, London Health Sciences Centre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sadeghirad B, Dodsworth BT, Schmutz Gelsomino N, Goettel N, Spence J, Buchan TA, Crandon HN, Baneshi MR, Pol RA, Brattinga B, Park UJ, Terashima M, Banning LBD, Van Leeuwen BL, Neerland BE, Chuan A, Martinez FT, Van Vugt JLA, Rampersaud YR, Hatakeyama S, Di Stasio E, Milisen K, Van Grootven B, van der Laan L, Thomson Mangnall L, Goodlin SJ, Lungeanu D, Denhaerynck K, Dhakharia V, Sampson EL, Zywiel MG, Falco L, Nguyen AV, Moss SJ, Krewulak KD, Jaworska N, Plotnikoff K, Kotteduwa-Jayawarden S, Sandarage R, Busse JW, Mbuagbaw L. Perioperative Factors Associated With Postoperative Delirium in Patients Undergoing Noncardiac Surgery: An Individual Patient Data Meta-Analysis. JAMA Netw Open. 2023 Oct 2;6(10):e2337239. doi: 10.1001/jamanetworkopen.2023.37239. PMID 37819663
- [Background] Bickel H, Gradinger R, Kochs E, Forstl H. High risk of cognitive and functional decline after postoperative delirium. A three-year prospective study. Dement Geriatr Cogn Disord. 2008;26(1):26-31. doi: 10.1159/000140804. Epub 2008 Jun 24. PMID 18577850
- [Background] Lawson RA, McDonald C, Burn DJ. Defining delirium in idiopathic Parkinson's disease: A systematic review. Parkinsonism Relat Disord. 2019 Jul;64:29-39. doi: 10.1016/j.parkreldis.2018.09.025. Epub 2018 Sep 26. PMID 30279060
- [Background] Lawson RA, Richardson SJ, Yarnall AJ, Burn DJ, Allan LM. Identifying delirium in Parkinson disease: A pilot study. Int J Geriatr Psychiatry. 2020 May;35(5):547-552. doi: 10.1002/gps.5270. Epub 2020 Feb 7. PMID 31994774
- [Background] Carlson JD, Neumiller JJ, Swain LD, Mark J, McLeod P, Hirschauer J. Postoperative delirium in Parkinson's disease patients following deep brain stimulation surgery. J Clin Neurosci. 2014 Jul;21(7):1192-5. doi: 10.1016/j.jocn.2013.12.007. Epub 2014 Jan 2. PMID 24518269
- [Background] Tanaka M, Tani N, Maruo T, Oshino S, Hosomi K, Saitoh Y, Kishima H. Risk Factors for Postoperative Delirium After Deep Brain Stimulation Surgery for Parkinson Disease. World Neurosurg. 2018 Jun;114:e518-e523. doi: 10.1016/j.wneu.2018.03.021. Epub 2018 Mar 9. PMID 29530688
- [Background] Astalosch M, Mousavi M, Ribeiro LM, Schneider GH, Stuke H, Haufe S, Borchers F, Spies C, von Hofen-Hohloch J, Al-Fatly B, Ebersbach G, Franke C, Kuhn AA, Kubler-Weller D. Risk Factors for Postoperative Delirium Severity After Deep Brain Stimulation Surgery in Parkinson's Disease. J Parkinsons Dis. 2024;14(6):1175-1192. doi: 10.3233/JPD-230276. PMID 39058451
- [Background] Likhvantsev VV, Berikashvili LB, Smirnova AV, Polyakov PA, Yadgarov MY, Gracheva ND, Romanova OE, Abramova IS, Shemetova MM, Kuzovlev AN. Intraoperative electroencephalogram patterns as predictors of postoperative delirium in older patients: a systematic review and meta-analysis. Front Aging Neurosci. 2024 May 13;16:1386669. doi: 10.3389/fnagi.2024.1386669. eCollection 2024. PMID 38803541
- [Background] Kinoshita H, Saito J, Kushikata T, Oyama T, Takekawa D, Hashiba E, Sawa T, Hirota K. The Perioperative Frontal Relative Ratio of the Alpha Power of Electroencephalography for Predicting Postoperative Delirium After Highly Invasive Surgery: A Prospective Observational Study. Anesth Analg. 2023 Dec 1;137(6):1279-1288. doi: 10.1213/ANE.0000000000006424. Epub 2023 Mar 14. PMID 36917508
- [Background] Serrano-Duenas M, Bleda MJ. Delirium in Parkinson's disease patients. a five-year follow-up study. Parkinsonism Relat Disord. 2005 Sep;11(6):387-92. doi: 10.1016/j.parkreldis.2005.05.002. PMID 16111911
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918